CLINICAL TRIAL: NCT01201213
Title: Median Effective Concentration of Bupivacaine, Levobupivacaine and Ropivacaine After Intrathecal and Extradural Injection for Pain Relief in the First Stage of Labour
Brief Title: Bupivacaine, Levobupivacaine and Ropivacaine After Intrathecal and Extradural Injection in Labour
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Audit pre regulatory inspection
Sponsor: NHS Tayside (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007AN01
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Pain
Keywords: Bupivacaine; levobupivacaine; ropivacaine
MeSH Terms: conditions — Pain | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Extradural bupivacaine (Active Comparator): Local anesthetic
  Interventions: Drug: local anaesthetic injection
- Extradural levobupivacaine (Active Comparator): local anaesthetic
  Interventions: Drug: local anaesthetic injection
- Extradural ropivacaine (Active Comparator): local anaesthetic
  Interventions: Drug: local anaesthetic injection
- Intrathecal bupivacaine (Active Comparator): local anaesthetic
  Interventions: Drug: local anaesthetic injection
- Intrathecal levobupivacaine (Active Comparator): local anaesthetic
  Interventions: Drug: local anaesthetic injection
- Intrathecal ropivacaine (Active Comparator): local anesthetic
  Interventions: Drug: local anaesthetic injection

INTERVENTIONS:
Drug: local anaesthetic injection — Single bolus of drug for pain relief in early labour

SUMMARY:
A need exists to define the best local anesthetic and technique for pain relief in early labour. We suggest that calculating the molar Median Effective Dose for bupivacaine, levobupivacaine and ropivacaine given both by the intrathecal (as a combined spinal epidural and epidural routes) would provide a valid comparison between the pain relieving properties of all three drugs, from which a reasoned assessment of side effects can be made.

DETAILED DESCRIPTION:
Despite 40 years of epidural analgesia, a consensus still does not exist regarding the best local anesthetic or the best technique for the provision of pain relief in early labour. Two new local anesthetics, levobupivacaine and ropivacaine, have recently been introduced into clinical practice because they have shown reductions in cardiovascular and cerebrovascular toxicity in several small animal, large animal and human volunteer studies. Evidence of improved safety from these studies suggest that the new local anesthetics should be used for surgical anesthesia, such as cesarean section, and limb block, where large volume, high concentrations of local anesthetics are required, and the risk of toxicity is high.

In contrast, the use of levobupivacaine and ropivacaine in small doses for analgesia in labour remains controversial, and bupivacaine remains the intrathecal and extradural local anesthetic of choice in many obstetric units. A change from bupivacaine to one of the newer drugs for analgesia in labour would require evidence documenting a distinct advantage of one the new local anesthetics in providing equivalent pain relief, but with less side effects.

Until now, intrathecal and epidural studies investigating the efficacy of bupivacaine, levobupivacaine and ropivacaine in obstetric anesthesia have focused on a comparison of % weight/volume solutions. However, close scrutiny of the chemical composition of local anaesthetics with the same % weight/volume shows marked differences in molar concentration.

The reason for differences in molar concentration are two-fold. Levobupivacaine is presented commercially as a base and not as a hydrochloride and therefore has 12.7% more molecules than the equivalent concentration of bupivacaine. In addition, ropivacaine has a smaller molecular weight than either drug and thus has 4.5% more molecules than bupivacaine and 8.4% less molecules than levobupivacaine. Although molar differences between drugs are relatively slight, a small reduction in molar concentration may provide similar pain relief, but result in a large reduction in side effects due to the shape and position of the efficacy and side effect dose response curves.

Comparative studies of all three drugs have been inconclusive. Intrathecal studies have shown a potency hierarchy of bupivacaine > levobupivacaine > ropivacaine, but equivalent potency between levobupivacaine and ropivacaine when injected with the opioid, sufentanil.

Epidural studies have also shown the potency of levobupivacaine to be equivalent or greater than ropivacaine, but, when combined with sufentanil at "equipotent doses", both have shown a longer duration of analgesia than bupivacaine.

Use of %w/v solutions, addition of opioids, pre-study assumptions of "equipotency" and variable definitions of pain relief have all served to confuse the issue of local anaesthetic potency and no definite conclusion exists as to whether any drug displays an advantage when given by either the intrathecal or epidural route.

A second controversy concerns the mode of drug administration. Although epidural analgesia is popular in Scotland for initiating pain relief in labour, major centres in the South of England, Europe and North America use a combined technique of spinal followed by epidural analgesia. The principal advantage is quicker pain relief, but the rapid onset of action may be associated with hypotension, motor block and technical failure.

A need exists to define the best local anesthetic and technique for pain relief in early labour. We suggest that calculating the molar Effective Dose for bupivacaine, levobupivacaine and ropivacaine given both by the intrathecal and epidural routes would provide a valid comparison between the pain relieving properties of all three drugs, from which a reasoned assessment of side effects could be made.

Thus, our aim is to compare molar concentrations of bupivacaine, levobupivacaine and ropivacaine when injected into the intrathecal and epidural spaces for pain relief in the first stage of labour, allowing a rational, molar comparison of the intrathecal and epidural efficacy of all three drugs, and thus providing a meaningful side effect profile. Only then can an informed decision be made regarding best practice.

Study design Phase IV, single centre, randomised, single-blind study in pain relief during early labor.

Primary objective To determine the median effective concentration of bupivacaine, levobupivacaine and ropivacaine after intrathecal and extradural injection for pain relief in the first stage of labor.

Secondary objectives To chart a derived dose response curve for bupivacaine, levobupivacaine and ropivacaine after intrathecal and extradural injection Determine the intrathecal / epidural potency ratio of each drug To measure the degree of motor block using Bromage and Straight Leg Raising scales To measure side effects such as hypotension, nausea and vomiting To measure mode of delivery and fetal outcome

Number and type of patients 162 patients requesting pain epidural relief in early labour

Recruitment and allocation All patients presenting to the ante natal clinic and not scheduled for cesarean section will be approached for recruitment to this study. Patients expressing an interest in participation will be given an information sheet and a written consent form. Patients will be given at least 24 hours to make a decision about study involvement. Allocation to six groups will be by computer randomised number generation.

Recruitment and allocation All patients presenting to the ante natal clinic and not scheduled for cesarean section will be approached for recruitment to this study. Patients expressing an interest in participation will be given an information sheet and a written consent form. Patients will be given at least 24 hours to make a decision about study involvement. Allocation to six groups will be by computer randomised number generation.

Inclusion criteria

* The patient is aged > 18 years
* The patient is in early labour ≤ 5cm cervical dilation
* The patient is American Association of Anaesthesiologists Grade I - II
* The patient provides written informed consent to participate in the trial prior to surgery.

Exclusion criteria

* The patient has any known chronic medical condition for which regular medication is required
* The patient has received any investigational drug within the 90 days prior to the study or is scheduled to receive one during the study period.
* The patient is scheduled for caesarean section
* The patient has received opioids in the last 4 hours
* The patient has evidence of alcohol or drug abuse
* There is evidence of obstetric complications
* The fetus has shown signs of intrauterine growth retardation
* The patient has findings on pre-study evaluations (e.g. laboratory results, medical history, physical examination, ECG) that are clinically significant in the investigator's opinion such to exclude entry into the study.

Intervention

Following informed and written consent, patients will be randomised into six groups:

Patients, ward staff and primary investigator will be blinded to the study drug. Study drugs will be prepared according to Hospital Department of Pharmacy guidelines on the preparation of drugs for clinical studies. All study preparations will be coded with an equal chance of receiving one of six infusions.

All patients will receive:

* Size 16g intravenous cannula
* Hartmann's solution 500ml infused at 100ml h-1
* Epidural analgesia or intrathecal analgesia in order to standardise the intervention

  3ml intrathecal starting at a mass of 10 µmol bupivacaine, levobupivacaine or ropivacaine by a combined spinal-epidural analgesia technique (groups A, B, C).

  o 20 ml epidural starting at a mass of 50 µmol bupivacaine, levobupivacaine or ropivacaine (groups D, E, F),

Intrathecal saline placebo will not be used because intrathecal injection influences subsequent epidural spread and increases the risk of hypotension.

Assessments The primary pain assessment will be the 100mm Visual Analog Scale. The visual analog will be performed pre-epidural, and at 5 minute intervals after epidural insertion for 30 minutes, and every 5 minutes for a further 15 minutes in "unsuccessful" patients as highlighted below.

Three responses to epidural analgesia will be charted.

1. Successful "Excellent"pain relief ≤ 10 mm at any time within 30 min of epidural insertion
2. Unsuccessful "Good or reasonable" pain relief > 10mm at all times within 30 min of epidural insertion, but ≤ 10 mm within 45min after rescue injection of 10ml 0.25% bupivacaine
3. Technical failure > 10mm at all times within 30 min of epidural insertion, and still > 10 mm within 45min despite rescue injection of 10ml 0.25% bupivacaine

Three decisions will be made based on each response:

Response

1. "Excellent"pain relief. Next patient receives: 1 mmol less intrathecal or 5 mmol less epidural local anaesthetic
2. "Good or reasonable" pain relief. Next patient receives: 1 mmol more intrathecal or 5 mmol more epidural local anaesthetic
3. Technical failure Next patient receives same mass of drug

Concomitant Medication Additional analgesia will be allowed only in accordance with this protocol. The patient will be allowed to take her present analgesic medication up to 12 hours preoperatively. Opiate-containing medication (including codeine containing combinations) will not be allowed less than 4 hours pre-study.

Statistical analysis Data analysis will proceed according to guidelines for randomised controlled trials. The first stage of analysis will be to use descriptive statistics to describe recruited individuals in relation to those eligible, and to investigate comparability of the trial arms at baseline. The primary analysis will be an intention-to-treat comparison between the two groups for both primary and secondary outcomes. The primary outcome will be presented as Effective Dose with confidence intervals. Categorical data will be presented as number and % of events.

Justification of sample size Two-way analysis with 6 groups. However the maximum number of logical comparisons within an effect can be reduced to 6 such that the threshold P value for significance at the P<0.05 level will be P=0.0085

The coefficient of variation from the isobole study is approximately 20%. The coefficient of variation from the an intrathecal study ranged from about 15% to 18%.

So to detect a nominal 30% difference in potency, we will need N=27 per group for an up-down design with 90% power.

Ethical Considerations:

This study will be conducted in accordance with the Declaration of Helsinki and the Guidelines on Good Clinical Practice. The study will be submitted to a Multi-Centre Research Ethics Committee followed by Local Research Ethics Committees for approval prior to commencing the study.

Safety Evaluation:

Side effects or adverse events. Assessments of blood pressure, respiratory rate, nausea, retching/vomiting and sedation at will occur at 5 minute intervals for the first 30 minutes after insertion of the epidural catheter, then at 45 minutes if necessary. The incidence and severity of nausea /vomiting/sedation will be assessed using a verbal rating score.

Serious Adverse Events will be defined as foetal or maternal haemodynamic or cerebral side effects occurring within 15 minutes of epidural or spinal injection

* Foetal heart rate < 100 bpm
* Maternal hypotension < 30% pre-epidural level
* Bradycardia <50bpm
* Any cardiac arrythmia
* Convulsions
* Residual neurological damage
* Dizziness or headache
* Fever > 38 centigrade

All serious adverse events will be immediately reported to the Ethics committee and Medicine and Health Regulatory Authority

ELIGIBILITY:
Inclusion Criteria:

* The patient is aged > 18 years
* The patient is in early labour ≤ 5cm cervical dilatation
* The patient is American Association of Anaesthesiologists Grade I - II
* The patient provides written informed consent to participate in the trial prior to surgery

Exclusion Criteria:

* The patient has any known chronic medical condition for which regular medication is required
* The patient has received any investigational drug within the 90 days prior to the study or is scheduled to receive one during the study period
* The patient is scheduled for caesarean section
* The patient has received opioids in the last 4 hours
* The patient has evidence of alcohol or drug abuse
* There is evidence of obstetric complications
* The fetus has shown signs of intrauterine growth retardation
* The patient has findings on pre-study evaluations (e.g. laboratory results, medical history, physical examination, ECG) that are clinically significant in the investigator's opinion such to exclude entry into the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Visual analogue pain score at 30minutes after epidural injection | 30 minutes
  To determine the median effective concentration of bupivacaine, levobupivacaine and ropivacaine after intrathecal and extradural injection for pain relief in the first stage of labour.

SECONDARY OUTCOMES:
Motor block | 45 minutes
  To chart a derived dose response curve for bupivacaine, levobupivacaine and ropivacaine after intrathecal and extradural injection Determine the intrathecal / epidural potency ratio of each drug To measure the degree of motor block using Bromage and Straight Leg Raising scales To measure side effects such as hypotension, nausea and vomiting To measure mode of delivery and fetal outcome

CONTACTS AND LOCATIONS:
Overall Officials: Graeme A McLeod, MD FRCA, Principal Investigator — NHS Tayside
Locations (1):
- Ninewells Hospital & Medical School, Dundee, Tayside, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
study terminated